CLINICAL TRIAL: NCT00403286
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group, Dose-Finding Trial to Evaluate the Safety and Efficacy of Fluticasone Propionate Combined With Formoterol Fumarate in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Dose-Finding Study Evaluating Safety and Efficacy in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director Clinical Affairs, Dey, L.P.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191-076
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic; Obstructive; Pulmonary; Disease; COPD; Safety; Efficacy; Pharmacokinetic; Dose-finding
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Disease | interventions — Fluticasone; Formoterol Fumarate; Fluticasone-Salmeterol Drug Combination

ARMS (8):
- C 10/1 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Formoterol Fumarate
- C 5/2 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Formoterol Fumarate
- C 5/1 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Formoterol Fumarate
- FP 1000 (Experimental)
  Interventions: Drug: Fluticasone Propionate
- FF 20 (Experimental)
  Interventions: Drug: Formoterol Fumarate
- AD 250/50 (Active Comparator)
  Interventions: Drug: Fluticasone Propionate/Salmeterol Xinafoate
- Plc (Placebo Comparator)
  Interventions: Drug: Placebo
- C 10/2 (Experimental)
  Interventions: Drug: Fluticasone Propionate/Formoterol Fumarate

INTERVENTIONS:
Drug: Fluticasone Propionate/Formoterol Fumarate — Inhalation suspension for nebulization 1000/20 mcg bid for 2 weeks
  Arms: C 10/2
Drug: Fluticasone Propionate/Formoterol Fumarate — Inhalation Suspension for nebulization 1000/10 mcg bid for 2 weeks
  Arms: C 10/1
Drug: Fluticasone Propionate/Formoterol Fumarate — Inhalation Suspension for nebulization 500/20 mcg bid for 2 weeks
  Arms: C 5/2
Drug: Fluticasone Propionate/Formoterol Fumarate — Inhalation Suspension for nebulization 500/10 mcg bid for 2 weeks
  Arms: C 5/1
Drug: Fluticasone Propionate — Inhalation Suspension for nebulization 1000 mcg bid for 2 weeks
  Arms: FP 1000
Drug: Formoterol Fumarate — Inhalation Solution for nebulization 20 mcg bid for 2 weeks
  Arms: FF 20
Drug: Fluticasone Propionate/Salmeterol Xinafoate — Inhalation Powder delivered by Diskus device 250/50 mcg bid for 2 weeks
  Arms: AD 250/50
Drug: Placebo — Inhalation Solution for nebulization 2 mL bid for 2 weeks
  Arms: Plc

SUMMARY:
The purpose of the study is to determine the appropriate dose of fluticasone propionate/formoterol fumarate that is closest to Advair Diskus (fluticasone propionate/salmeterol xinafoate using pulmonary function, safety, and levels of study drug in blood plasma in patients with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Female of child-bearing potential to use adequate birth control
* Smoker or ex-smoker with history of at least 10 years of smoking at least one pack of cigarettes per day
* Meet lung function requirements

Exclusion Criteria:

* Diagnosis of asthma
* Other significant disease than COPD
* Pregnant or lactating female
* Female planning to become pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
2-hour post-dose FEV1 | 2 weeks
AUC(0-12) and Cmax in plasma | 2 weeks
pre-dose FEV1 | 2 weeks
Amount and percent total dose excreted in urine | 2 weeks

SECONDARY OUTCOMES:
FEV1 AUC(0-2) | 2 weeks
COPD exacerbations
Treatment Emergent Adverse Events | 2 weeks

CONTACTS AND LOCATIONS:
Locations (47):
- United States (47):
  - Research Site, Birmingham, Alabama
  - Research Site, Jasper, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Buena Park, California
  - Research Site, Costa Mesa, California
  - Research Site, Encinitas, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Tamarac, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Hines, Illinois
  - Research Site, Lenexa, Kansas
  - Research Site, Topeka, Kansas
  - Research Site, Madisonville, Kentucky
  - Research Site, Wheaton, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, Cherry Hill, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Camillus, New York
  - Research Site, Liverpool, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Morrisville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, East Providence, Rhode Island
  - Research Site, Spartanburg, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, South Burlington, Vermont
  - Research Site, Abingdon, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin